CLINICAL TRIAL: NCT00100243
Title: Phase 2 Study of Abarelix in Androgen-Independent Prostate Cancer Progressing After Agonist Therapy
Brief Title: Study of Abarelix in Androgen-Independent Prostate Cancer Progressing After Agonist Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PRAECIS Pharmaceuticals Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 149-04-01
Record Dates: First submitted 2004-12-27; First posted 2004-12-28 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Prostate Cancer
Keywords: androgen-independent; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abarelix

INTERVENTIONS:
Drug: Plenaxis

SUMMARY:
This is a Phase 2, open-label study in subjects with androgen-independent prostate cancer who have progressed following treatment with an LHRH agonist. Up to 22 subjects will be enrolled. Enrollment will be monitored to ensure that not all subjects are enrolled based on rising prostate specific antigen (PSA) criterion only.

Subjects will be treated with abarelix (Plenaxis) 100 mg intramuscularly (IM) every 2 weeks for 12 weeks (total dose of 600 mg).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histologically or cytologically confirmed prostate cancer that has progressed within 60 days of the start of screening despite castrate levels of testosterone from treatment with an LHRH agonist. Progression will be defined as one or more of the following: *A rising PSA, defined as at least two consecutive rises in PSA over a reference value (PSA #1). The first rising PSA (PSA #2) must be taken at least one week after PSA #1. A third PSA (PSA #3) is required to be greater than PSA #2; if not, a fourth PSA (PSA #4) is required to be greater than PSA #2, OR

  * The appearance of new metastatic lesions on a bone scan, OR
  * Progression of known lesions or the appearance of new metastatic lesions on CT, MRI, chest x-ray, or other radiographic evaluations.
* Subject whose hormonal therapy includes an anti-androgen must have the anti-androgen discontinued prior to the start of screening (at least 6 weeks for bicalutamide and at least 4 weeks otherwise). If there is a reduction in the PSA after anti-androgen withdrawal, the subject must continue to demonstrate progression as defined above after anti- androgen withdrawal to be eligible.
* ECOG Performance Status ≤ 3
* Age ≥ 18 years of age
* Life expectancy ≥ 6 months
* Serum testosterone less than or equal to 50 ng/dL
* PSA ≥ 5 ng/mL (if progression is determined from a rise in PSA)
* WBC greater than or equal to 3,000/mm3
* Hematocrit ≥ 30%
* Platelet count greater than or equal to 100,000/mm3
* Serum creatinine less than or equal to 2 x upper limit of normal (ULN)
* Bilirubin (direct or total) less than or equal to 2 x ULN
* SGPT (ALT) and SGOT (AST) less than or equal to 2 x ULN

Exclusion Criteria:

A subject is ineligible to participate in the study if he meets any of the following criteria:

* Prior treatment for prostate cancer with:

  * Chemotherapy
  * Radiopharmaceutical such as strontium or samarium
  * Diethylstilbesterol or another estrogen agonist or antagonist
  * Ketoconazole
  * Aminoglutethimide
* Current treatment with Class IA (e.g., quinidine, procainamide) or Class III (e.g., amiodarone, sotalol) antiarrhythmic medication
* Currently taking PC SPES
* History of allergy to a LHRH agonist or GnRH antagonist
* Major surgery within 4 weeks
* Serious medical illnesses, including malnutrition, that in the judgment of the investigator would preclude protocol treatment
* Significant cardiovascular illness defined as NYHA class III or IV congestive heart failure or unstable angina within 6 months, myocardial infarction within 12 months, deep venous thrombosis within 2 years, or any history of acute pulmonary embolism
* Active second malignancy other than non-melanoma skin cancer or superficial bladder cancer
* Any uncontrolled infection, including HIV
* Any other experimental therapy within 4 weeks prior to study entry
* QTc > 450 msec on a screening ECG obtained by the investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2004-05; Study Completion 2005-09

PRIMARY OUTCOMES:
Clinical adverse events, laboratory abnormalities, and withdrawals due to adverse events
Serum FSH levels below the lower limit of quantitation (LLOQ) on Days 57 and 85

CONTACTS AND LOCATIONS:
Overall Officials: Marc Garnick, MD, Study Director — PRAECIS Pharmaceuticals Inc.
Locations (7):
- United States (7):
  - San Diego Center for Urology, La Mesa, California
  - Southwest Florida Urological Associates, Fort Myers, Florida
  - Panama City Urological Center, Panama City, Florida
  - Columbus Urology Research, LLC, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina